CLINICAL TRIAL: NCT02102958
Title: Nonvisual Foot Examination for People With Diabetes and Visual Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R21NR012513 (NIH)
Record Dates: First submitted 2014-03-31; First posted 2014-04-03 (Estimated); Last update posted 2023-11-14 (Actual); Status verified 2014-03

CONDITIONS: Diabetes; Visual Impairment
Keywords: diabetes; visual impairment; foot care; diabetes self-management education
MeSH Terms: conditions — Diabetes Mellitus; Vision Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental (Experimental): DSME with Nonvisual Foot Examination
  Interventions: Behavioral: DSME with Nonvisual Foot Examination
- Comparison (Active Comparator): DSME with Usual Foot Examination Instruction
  Interventions: Behavioral: DSME with Usual Foot Examination Instruction

INTERVENTIONS:
Behavioral: DSME with Nonvisual Foot Examination — Diabetes Self-Management Education (DSME) with Nonvisual Foot Examination included comprehensive DSME taught by Certified Diabetes Educators that included instruction in nonvisual self-examination of feet using the senses of touch and smell.
  Arms: Experimental
Behavioral: DSME with Usual Foot Examination Instruction — DSME with usual foot examination instruction was comprehensive diabetes self management education taught by Certified Diabetes Educators that included usual care instructions for examination for feet at home by visually impaired persons, i.e., to have a sighted person check the feet regularly.
  Arms: Comparison

SUMMARY:
Because people who have both diabetes and visual impairment have high risk for foot problems, prevention of ulcers and amputation is a high priority. Usual care in diabetes self-management education (DSME) is to teach them to seek sighted assistance for regular foot examination, yet clinical experience suggests that this advice is seldom heeded. One possible solution is to teach use of the nonvisual senses of touch and smell for a systematic, thorough foot self-examination. The purpose of this pilot study was to compare the efficacy, acceptability, and feasibility of nonvisual foot examination with usual care (examination of the visually impaired person's feet by a sighted family member or friend).

ELIGIBILITY:
Inclusion Criteria:

* over age 18
* diagnosed with either type 1 or type 2 diabetes
* stated they had visual impairment

Exclusion Criteria:

* unable to pass a brief decisional capacity test
* had a score above 80 on the near vision scale of the National Eye Institute Visual Functioning Questionnaire
* had bilateral lower extremity amputations
* by self-report were unable to sense light touch on two or more fingers or either hand

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2011-07; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Frequency of foot examination at home | 6 months
  number of times that the enrolled participant or someone else examined the person's feet at home during the study period

SECONDARY OUTCOMES:
New foot problems discovered at home | 6 months
  total number of new foot problems reported to podiatrists as having been discovered at home by the participant or someone else examining the person's feet

OTHER OUTCOMES:
Total new foot problems | 6 months
  total number of foot problems documented by the podiatrist at podiatry visit

CONTACTS AND LOCATIONS:
Overall Officials: Ann S Williams, PhD, Principal Investigator — Case Western Reserve University
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States